CLINICAL TRIAL: NCT07026240
Title: Post-operative Monitoring of Gastric Cancer Using Circulating DNA in Blood Samples
Brief Title: Post-operative Monitoring of Gastric Cancer
Status: Recruiting | Type: Observational
Sponsor: Suzhou Huhu Health & Technology Inc. (Industry)
Collaborators: Fudan University (Other)
Responsible Party: Sponsor
Other Study IDs: 2311285-6（1）
Record Dates: First submitted 2025-06-04; First posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Human Papillomavirus DNA Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood samples collected from each study participant.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- malignant group: Subjects diagnosed with gastric cancer.
  Interventions: Diagnostic Test: DNA test

INTERVENTIONS:
Diagnostic Test: DNA test — a new non-invasive detection method for postoperative monitoring of gastric cancer in the blood

SUMMARY:
This study is to determine the performance of non-invasive new multi-target biomarkers in the post-operative monitoring of gastric cancer.

DETAILED DESCRIPTION:
This study aims to develop and validate a new non-invasive detection method for postoperative monitoring of gastric cancer in the blood. Blood will also be collected at various time points post-operatively. We will determine whether these new biomarkers can be used as prognostic biomarkers to predict tumor recurrence and metastasis. We will also determine whether these new biomarkers detect tumor recurrence and metastasis earlier than methods currently used in the clinic such as imaging and tumor biomarkers CA19-9, CEA, and CA72-4.

This study is a prospective and multi-center study.

ELIGIBILITY:
Inclusion Criteria:

1. Subject age over 18.
2. Subject has stomach discomfort, and seek medical attention at the Gastric Surgery Department of our center.
3. Subject has or will have gastroscopy and/or pathological examination results at this center.
4. Subject must be able to fully understand the informed consent form and be able to personally sign it.

Exclusion Criteria:

1. Subject has serious heart, liver, kidney dysfunction, or mental illness.
2. Subject diagnosed previously with any kind of malignant tumor.
3. Subject is known to be infected with HIV or other related diseases (considering interference from the use of immune drugs).
4. Subject is receiving targeted drugs, immunosuppressants, immunomodulators, and biological therapies.
5. Researchers believe that subject is not suitable for enrollment.
6. Subject can not supply sufficient sample to complete this experiment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects age over 18, regardless of gender or region, and those who meet the inclusion criteria for this clinical trial, are eligible to enroll at the designated clinical sites. More than 258 subjects are targeted to enroll.
Sampling Method: Non-Probability Sample
Enrollment: 258 (Estimated)
Dates: Start 2024-02-18 (Actual); Primary Completion 2026-01-07 (Estimated); Study Completion 2026-01-07 (Estimated)

PRIMARY OUTCOMES:
The performance of the new biomarkers in the post-operative monitoring of gastric cancer | 2 years
  Number of Participants With Tumor Recurrence Detected by the New System vs. Imaging and Serum Markers (CA19-9, CEA, CA72-4).

SECONDARY OUTCOMES:
Metastasis Detection Time: New vs. Conventional Methods | 2 years
  Time to Detection of Metastasis (Days) by the New System Compared to Conventional Methods.

CONTACTS AND LOCATIONS:
Overall Officials: Dazhi Xu, MD., PhD,, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No